CLINICAL TRIAL: NCT04935905
Title: Accuracy of Peak Cough Flow Measurements Using a Mechanical Insufflator-exsufflator in Patients With Neuromuscular Disease: A Single Centre Prospective Observational Study
Brief Title: Accuracy of Peak Cough Flow Measurements Using a Mechanical Insufflator-exsufflator
Acronym: MIEPCF
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 272851
Record Dates: First submitted 2020-02-05; First posted 2021-06-23 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical Insufflator-Exsufflator — This device augments a cough by applying a positive pressure via the upper airway or tracheostomy to increase lung volume to maximal inspiratory capacity, followed by a rapid and quick change to negative pressure to increase expiratory flow and simulate normal cough mechanism

SUMMARY:
The primary aim of this study is to evaluate the agreement of MIE devices measurement of MIE assisted peak cough flow (PCF) compared with a pneumotachographs during usual MIE care. This will be the first study to do this through range of MIE pressures and include patients who are receiving MIE via a tracheostomy. It will also aim to evaluate the intra-subject repeatability of measures for patients who receive more than one MIE cycle as part of their usual care. It will be the first to measure MIE assisted PCF contemporaneously during intervention using the gold standard pneumotachograph. This will inform treatment effect size and the efficacy of usual practice MIE in augmenting PCF measurements above critical cut off values for effective cough and secretion clearance.

Finally the study will also aim to understand how patients perceive the impact of MIE in clearing secretions from their chest by asking them to rate presence of chest secretions pre and post intervention using a visual analogue scale (VAS)

DETAILED DESCRIPTION:
Patients with a neuromuscular disease (NMD) lose strength in their breathing muscles which leads to an inability to generate an effective cough. Peak Cough Flow (PCF) is a simple objective measure of cough and is the recommended measure in patients with NMD. Critical peak cough flow values are used to evaluate cough, these include PCF less than 160 L/min to indicate an ineffective cough, PCF between 161- 270 to indicate an impaired cough and PCF greater than 270 L/min to indicate an effective cough. Mechanical insufflator- exsufflator (MIE) devices more commonly known as 'cough assist' devices have an inbuilt measure of PCF however they aren't currently recommended for use to due to limited information available regarding their accuracy. This will be a single centre prospective observational study. Once patients have consented to participate in the study, they will be visited once on the unit during their admission by the researcher with the visit lasting approximately an hour.

During the visit they will receive their usual care MIE with a pneumotachograph fitted into the circuit. The primary outcome is the agreement of MIE assisted PCF measures between the MIE device and pneumotachograph. Before and after the intervention the patient will be asked to rate the presence of mucous in their lungs using a visual analogue scale.

The following data will be recorded

* Neuromuscular diagnosis
* Age, height, weight,
* Comorbidities
* Hospital length of stay (Days)
* Ventilation dependency(hours/Day)
* Bronchodilator and/or mucolytic medications
* Vital observations (heart rate, blood pressure, oxygen saturations)
* Method of MIE delivery (mask or tracheostomy)
* Tracheostomy size, type and brand
* Bulbar function if available (Laryngoscope)
* Spirometry - Forced Expired Volume in 1 second (FEV1), Forced Vital Capacity (FVC), (from clinical notes)
* Voluntary PCF (collected from patient by researcher)
* MIE Mode (collected from device by researcher)
* MIE Total number cycle repeats (collected from device by researcher)
* MIE device Inspiratory pressure (collected from device by researcher)
* MIE inspiratory pressure at interface (Pressure transducer)
* MIE inspiratory time (collected from device by researcher)
* MIE peak inspiratory Flow (from device by researcher)
* MIE device expiratory pressure (collected from device by researcher)
* MIE expiratory pressure at interface (Pressure transducer)
* MIE Expiratory time (collected from device by researcher)
* MIE Assisted PCF Pneumotachograph (From patient by researcher)
* MIE Assisted PCF MIE (From patient by researcher)
* Visual Analogue Scale regarding secretion presence pre and post MIE (from patient by researcher)

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuromuscular disease-related respiratory failure and are receiving MIE as part of their usual care
* Patients who are clinical stable and documented as such by the supervising clinician
* Patients who are cognitively intact and have the capacity able to provide informed consent

Exclusion Criteria:

* Pregnancy
* Aged <18
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient with neuromuscular related respiratory failure and receiving MIE as part of their usual care
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Agreement of Peak Cough Flow between MIE and pneumotachograph. | Data will be collected at the point of recruitment to the study and then be reported within 1 year
  Peak Cough Flow measure the peak flow of expired air during the exsufflation phase of cough or MIE assisted cough

SECONDARY OUTCOMES:
Visual Analogue Scale | Data will be collected at the point of recruitment to the study and then be reported within 1 year
  Patients will be asked regarding their perceived presence of chest secretions pre and post and post intervention using the visual analogue scale. The scale ranges from 0 to 10 with 10 being the highest perceived score.
Treatment effect size of PCF during usual MIE care | Data will be collected at the point of recruitment to the study and then be reported within 1 year
  Will compared baseline voluntary PCF to MIE assisted PCF
Exploratory analysis of MIE Pressure and PCF | Data will be collected at the point of recruitment to the study and then be reported within 1 year
  Exploratory analysis of the correlation between MIE Pressure with PCF and cough function will be performed using chi square, correlation and logistic regression as appropriate.
Exploratory analysis of MIE inspiratory Volume and PCF | Data will be collected at the point of recruitment to the study and then be reported within 1 year
  Exploratory analysis of the correlation between MIE inspiratory volume with PCF and cough function will be performed using chi square, correlation and logistic regression as appropriate.
Intra-subject variance of repeated PCF measures | Data will be collected at the point of recruitment to the study and then be reported within 1 year
  For patient receiving more than one cycle of MIE during their usual care, the repeated PCF measures taken by MIE and Pneumotachograph and variance of measures evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Osman, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St. Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided